CLINICAL TRIAL: NCT00624000
Title: IV vs. IA tPA (Activase) in Acute Ischemic Stroke With CTA Evidence of Major Vessel Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Susan Wilson, Sub-Investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB-IND # 11364
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tetradecanoylphorbol Acetate; Tissue Plasminogen Activator

ARMS (2):
- 1 (Experimental): IA administration of Alteplace vs. IV administration of Alteplace
  Interventions: Drug: IV tpa (Alteplase) vs IA tpa (Alteplase)
- 2 (Active Comparator): IA administration of Alteplase vs.IV administration of Alteplase
  Interventions: Drug: IV tpa (Alteplase) vs IA tpa (Alteplase)

INTERVENTIONS:
Drug: IV tpa (Alteplase) vs IA tpa (Alteplase) — Alteplase was administered Either IA or IV x 1

SUMMARY:
Stroke is the third leading cause of death in the United States, responsible for 158,488 deaths in 1998 (American Heart Association). Nationwide, each year, an estimated 600,000 to 750,000 people suffer a new or recurrent stroke. Cerebral infarction comprises 80% of all strokes and is the result of a complex series of cellular metabolic events that occur rapidly after interruption of blood flow to a region of the brain. The extent of the brain damage is dependent on the duration and severity of the cerebral ischemia. Acute thrombus formation or migration is the principal cause of blood flow interruption in at least 75% of cerebral infarctions. In several animal models of focal cerebral ischemia, restoration of cerebral blood flow within two to six hours after initial occlusion has been associated with smaller volumes of cerebral infarction and improved functional outcome. An effective way of dissolving the thrombus is by administration of recombinant tissue plasminogen activator or Activase (Alteplase, rt-PA), which promotes the proteolytic action of plasmin from plasminogen at the site of a clot. In this study, the drug, Activase, will be administered in subjects with acute ischemic stroke (AIS) intravenously (IV) or by local intra-arterial (IA) injection. The use of the intravenous administration within 3 hours of stroke symptom onset is FDA approved whereas the intra-arterial administration, despite evidence of potential benefit, is not currently FDA approved. Although not FDA approved, this study will evaluate the effectiveness of IA thrombolysis with Activase, used in AIS because of its higher rate of recanalization , potential expansion of the time window out to 6 hours, and lower doses of thrombolytic agent used compared with systemic or intravenous Activase. The study is designed to test the feasibility and provide preliminary safety data regarding the relative benefits and risks of IA Activase as compared to IV Activase when administered per the NINDS rt-PA stroke study protocol, i.e. randomized within 3 hours of onset of symptoms of ischemic stroke then treated within 3 hours in the IV Activase arm and within 4 hours in the IA Activase arm.

DETAILED DESCRIPTION:
DESCRIPTION OF THE STUDY This is a randomized, controlled, single center feasibility and preliminary safety study to determine the clinical efficacy of Activase administered locally, IA, in the course of an angiogram, as compared with Activase systemic IV infusion, in subjects with a ischemic stroke due to major vessel occlusion (M1, M2, terminal ICA, basilar or vertebral) detected by CT angiography, within 3 hours of symptoms onset. IV Activase (0.9 mg kg-1, maximum 90 mg) will be administered as per the NINDS protocol and IA Activase (2 mg bolus, followed by 10 mg hr-1 for 2 hours or TIMI 3 recanalization, whichever is earlier, maximum total dose 22 mg) will be administered as per the protocol used in the IMS-2 study with administration initiated within 4 hours from symptom onset and completed within 6 hours from symptom onset. The subject will be randomized following CT angiography after the demonstration of complete occlusion or minimal perfusion of symptom-related M1 segment and/or M2, distal ICA, vertebral artery or basilar artery. The primary analysis will be focused on feasibility of such a trial in terms of time-frame, preliminary safety analysis (the proportion of symptomatic intracranial hemorrhages) and preliminary risk-benefit ratio of IA Activase when compared with IV Activase. Secondary analyses will include the proportion of subjects exhibiting significant neurological improvement, reduction in disability and recanalization on a MRA or CTA. The sample size for this feasibility trial was estimated taking into account that it will be done in a single center, involve a major investment in time, personnel, and equipment required. IA thrombolysis as compared to IV thrombolysis, should be justified only with evidence of a superior clinical efficacy. A larger multicenter feasibility trial will need to be planned to determine safety and estimate sample size for an efficacy trial. An outside, independent safety monitor will assess the safety of the treatment arms.

A majority of clinical trials involving AIS conducted since the NINDS Activase stroke study have yielded negative results, emphasizing the point that recanalization and not neuroprotection can lead to clinical improvement. A recent randomized clinical trial (PROACT) showed the efficacy (recanalization and clinical improvement) of IA thrombolysis with Prourokinase for acute ischemic stroke <6 h from symptom onset, due to occlusion of proximal MCA. Although not FDA approved, IA thrombolysis with Activase, used in AIS is attractive because of higher rates of recanalization, potential extension of the time window out to 6 hours from symptom onset, and lower doses of thrombolytic agent used compared with systemic or IV Activase and a possible lower rate of symptomatic ICH (5-7%) compared with IA Pro-UK (10.9%). Support for use of IV Activase comes mainly from the NINDS study, whereas that for IA Activase comes from the PROACT study and a metanalysis of several anecdotal series. However, these two therapeutic approaches have never been compared in a randomized controlled trial. IA Activase may be used in AIS due to major vessel occlusion, whereas IV Activase may be used independent of the presence or absence of major vessel occlusion. CT angiography can rapidly detect major vessel occlusion and hence candidacy for IA thrombolysis. An ongoing pilot (IMS-2 trial) assessing the use of combination of IV and IA thrombolysis and comparing it with historical control has one draw-back in that the subjects are being subjected to a dual risk of hemorrhage by IV (6%) + IA (5-7%) Activase.

The rationale for the study design is as follows:

* Random assignment: to reduce treatment assignment bias.
* Controlled: the appropriate control group being the FDA approved IV Activase administration.
* Open label: as intra-arterial and intravenous administration is difficult to blind observers because of the difference in route of administration that is obvious to the observer and the subject. Sham intra-arterial stick that can be used to camouflage the information, may be extremely dangerous in the intra-venous group.
* Blinded 90-day assessment: to remove assessment bias.

Method of Treatment Assignment Block randomization (1:1) will be used to assign equal numbers of subjects to the IV and IA arms. In the preliminary feasibility study twelve subjects will be randomly assigned to receive IV (N=6) and IA (N=6) Activase. The treatment will remain open label to the treating physician. A physician blinded to the treatment arm will assess the 90-day outcomes.

Study Treatment Activase will be administered IV or IA based on random assignment. The IV administration will be in accordance to the FDA approved guidelines based on the NINDS rt-PA stroke study. The IA administration is considered investigational and will be in accordance to the ongoing IMS-2 study.

Cathetrization and Intra-arterial Alteplase protocol: A sheath will be placed in the femoral artery by a 1-wall puncture and arteriography performed by standard technique. If the suspected distribution of ischemia is the carotid artery, injection of the common carotid artery for examination of the carotid bifurcation as well as for intracranial examination will be performed. If the suspected arterial distribution is vertebral or basilar artery, selective injection of both vertebral arteries will be performed. Arteriographic examination of the remainder cerebral vessels will be performed if examination of collateral flow to the brain is deemed essential for determining treatment strategies. Five thousand units of heparin will be administered IV as a bolus at the beginning of the procedure. No post bolus IV heparin will be administered. Per standard neurointerventional procedure, a heparin flush solution (eg, 1000 U in 500 mL) normal saline at ~2 U of heparin/min) will be used through the access sheath and continued till the sheath is removed.

After performing diagnostic cerebral arteriogram, a 3F, tapered, variable-stiffness, end-hole microcatheter will be passed over a micro-guide wire to the level of occlusion. One milligram of Activase will be injected beyond the thrombus and the catheter retracted into the proximal thrombus where an additional one milligram of Activase will be injected. A maximum of 22 mg of Activase will be administered in pulse spray fashion at a rate of 1mg every 6 minutes up to 10 mg/hr for 2 hrs till the maximum dose is reached or a TIMI 3 flow is noted on arteriographic examination. Repeat arteriography will be performed every 15 minutes using isosmolar contrast during the intra-arterial administration to assess recanalization. If the vessel is not patent the intra-arterial administration is continued. If the vessel is partially recanalized, the infusion catheter is introduced further into the vessel for thrombus access. If the arterial catheter cannot be introduced into the thrombus, the Activase will be administered proximal to the thrombus as described above. The subject's neurological function will be evaluated every 15 minutes during the IA procedure, including level of consciousness, speech examination, cranial nerve examination, and upper extremity motor and sensory function.

If the subject did not have an occlusion on the initial arteriogram in the vascular territory appropriate for the subject's symptoms, no Activase will be administered, and the procedure terminated (these subjects will be included in the overall analysis). If the subject has a significant stenosis or occlusion of the internal carotid, vertebral or basilar arteries, the stenosis/occlusion is traversed with the microcatheter to approach a distal occlusive thrombus. The use of Activase(IV) in an acute ischemic stroke is standard of care. IA Activase is being performed clinically, but is not standard of care. Intravenous Activase protocol: is essentially identical to the NINDS rt-PA stroke study. In accordance with the protocol, AIS subjects will be treated with IV Activase within 180 minutes from symptom onset. Symptom onset is defined in the usual manner as the last time at which the subject was known to be asymptomatic. A total dose of 0.9 mg/kg body weight (max 90 mg) will be administered, 10% of it given as IV push over 1 minute and the remainder 90% as an IV infusion over 1 hour.

One week, one month, and three months after receiving Activase IV or IA the subject will spend 10 to 20 minutes talking to a doctor and being examined to check recovery from the stroke. In addition, 60 days after receiving the study drug, the study coordinator will contact the subject by phone to ask questions about overall feeling of health. This telephone contact is expected to take about five minutes. One follow-up visit after the subject has left the hospital is standard care for someone who has had a stroke. Other visits and the telephone call are for research purposes only.

Outcome Measures

Primary Efficacy Outcome Measures

The following primary efficacy outcome measures will be evaluated:

* Feasibility of enrolling 12 subjects with major vessel occlusion within 1 year and random 1:1 assignment to treatment with IV (N=6) and IA (N=6) IA Activase using the following criteria: - Time to clinical and radiological assessments

  * Time to IA Activase treatment
  * Proportion of subjects receiving timely assessments and treatment
* Preliminary safety assessment: 24 hour symptomatic ICH
* Resources utilized and risk-benefit of IA Activase treatment.

Secondary Outcome Measures

The following secondary efficacy outcome measures will be evaluated:

* 90-day efficacy outcome including NIHSS, modified Rankin Scale and Barthel's Index.
* 24-h recanalization (TIMI 2/3) on MRA or CTA
* Major extracranial bleed (defined under section 3.3.3) and asymptomatic intracranial hemorrhage

ELIGIBILITY:
Inclusion Criteria:Subjects will be eligible if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Age > 18 years
* NIHSS ≥ 4 or isolated aphasia or isolated hemianopsia

Exclusion Criteria:

* NIHSS >30
* Coma
* Rapidly improving symptoms
* History of stroke in the last 6 weeks
* Seizure at onset
* Subarachnoid Hemorrhage (SAH ) or suspected SAH
* Any history of Intracrannial Hemorrhage (ICH)
* Neoplasm
* Septic embolism
* Surgery, biopsy, trauma or LP in last 30 days
* Head trauma in the last 90 days
* Bleeding diathesis, or INR >1.7 or PTT >1.5 times baseline or platelet <100K
* SBP >180 or DBP ≥100 despite treatment with 3 doses of IV Labetalol (10-20 mg Q10")
* Lacunar stroke syndrome
* CT: Hemorrhage, tumor (except small meningioma), significant mass effect, midline shift, acute hypodensity or >1/3 MCA territory sulcal effacement
* Radiological contrast hypersensitivity
* Angiographic: Dissection, lack of access, lack of occlusion, or nonatherosclerotic arteriopathy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2004-03; Primary Completion 2007-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of enrolling 12 subjects with major vessel occlusion within 1 year and random 1:1 assignment to treatment with IV (N=6) and IA (N=6) IA Activase using the following criteria: Time to clinical and radiological assessments | 3 years
Time to IA Activase treatment | 3 years
Preliminary safety assessment: 24 hour symptomatic ICH | 3 years
Resources utilized and risk-benefit of IA Activase treatment. | 3 years

SECONDARY OUTCOMES:
90-day efficacy outcome including NIHSS, modified Rankin Scale and Barthel's Index. | 3 years
24-h recanalization (TIMI 2/3) on MRA or CTA | 3 years
Major extracranial bleed (defined under section 3.3.3) and asymptomatic intracranial hemorrhage. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Souvik Sen, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina Stroke Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Sen S, Huang DY, Akhavan O, Wilson S, Verro P, Solander S. IV vs. IA TPA in acute ischemic stroke with CT angiographic evidence of major vessel occlusion: a feasibility study. Neurocrit Care. 2009;11(1):76-81. doi: 10.1007/s12028-009-9204-1. Epub 2009 Mar 10. PMID 19277904